CLINICAL TRIAL: NCT03383536
Title: Social Withdrawal Following Trauma Exposure: a Neuroeconomic Approach
Brief Title: Neuroeconomics of Social Behavior Following Trauma Exposure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elizabeth Olson, Instructor, Mclean Hospital
Other Study IDs: 2017P001423; K23MH112873-01A1 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: fMRI; stress; peptide; social; neuroimaging
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for PACAP (stress peptide) analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase 1: Healthy control participants will provide neuroeconomic game responses to form a pool of potential responses for participants to interact with during Phase 2.
- Phase 2: PTS-SA: posttraumatic spectrum-socially anhedonic
- Phase 2: PTS-nonSA: posttraumatic spectrum-non-socially anhedonic
- Phase 2: HC: healthy controls

SUMMARY:
This study will use a neuroeconomic paradigm with state-of-the-art imaging protocols to probe abnormal social reward processing underlying social withdrawal in symptomatic trauma-exposed women. By also gathering self-report measures of social anhedonia, performance on non-social and social reward valuation tasks, and measures of real-world social functioning including social network size, we aim to specify how alterations in social reward processing result in social withdrawal and functional impairment.

DETAILED DESCRIPTION:
Impaired social functioning is a frequent and disabling sequela of trauma-related disorders. PTSD is associated with a high rate of severe impairment in quality of life relative to other anxiety disorders, including panic disorder, social phobia, and OCD, with particularly marked impairment in social quality of life. Mounting evidence indicates that impairment in quality of life in PTSD is strongly related to its effect on social functioning. Such difficulties are widespread and affect multiple social networks, including marital relationships, and friendships and family relationships. Social withdrawal, defined here in terms of reduced social network size, is of particular interest because of its strong relationship with health outcomes, including increased risk of disability, reduced immune response, and increased mortality risk; most critically, poor social integration is associated with a threefold increase in suicide risk. Because women are at a 2.3-to-3-fold increased risk compared to men of developing PTSD following trauma, understanding the differential neurobiological pathways that may contribute to the development of stress-related disorders in women is particularly critical. Women are more likely than men to endorse social detachment following trauma, especially when the trauma involves exposure to violence.

In this project, we propose abnormal reward processing (anhedonia) as a specific mechanism underlying social withdrawal in trauma-exposed women, and we present a paradigm that capitalizes on advances in neuroeconomics to elucidate the neural underpinnings of social withdrawal. Additionally, we propose to identify the possible influences of a stress peptide (pituitary adenylate cyclase-activating polypeptide: PACAP) implicated in sex-specific changes in social behavior following stress exposure.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Age 18-45
* Self-reported healthy volunteer status

Exclusion Criteria:

* Inability to provide written informed consent in English
* Inability to see task due to visual impairment
* Participants who produce T-scores of 65 or higher on any Brief Symptom Inventory (BSI) subscales will not be eligible to remain in the Trust Task participant pool.

Phase 2:

Inclusion Criteria:

* Female
* Trauma exposure appropriate to group
* For trauma-exposed groups the index trauma is actual or threatened physical assault or sexual violence
* PCL-5 score 33 and above (for PS-SA and PS-nonSA groups)
* Right handedness
* Age 18-45
* English as a first language

Exclusion Criteria:

* History of neurological illness (including head injury with loss of consciousness > 5 minutes)
* Medical conditions that may influence neuroimaging (e.g. HIV)
* Current or past DSM-5 Axis I disorder (for HC group)
* History of bipolar disorder or schizophrenia spectrum disorder
* Contraindications for MRI
* Alcohol dependence in the past 5 years
* Substance dependence in the past 3 years
* Daily substance use in the past year
* Prescribed psychotropic medication use in the past month
* Wechsler Abbreviated Scale of Intelligence- Second Edition (WASI-II) FSIQ < 70.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Phase 1 will include healthy volunteers (age 18-45, n = 60).
  Phase 2 will include posttraumatic spectrum-socially anhedonic women (PTS-SA, n = 36), posttraumatic spectrum-non-socially anhedonic women (PTS-nonSA), and healthy controls (HC, n = 36).
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Group differences in neuroeconomic game performance | Measured on the day of the MRI scan
  Compared to the PTS-nonSA and HC groups, the PTS-SA group will demonstrate lower investments and slower learning rates on the Trust Task than on the non-social risk task compared with PTS-nonSA and HC subjects
Group differences in fMRI BOLD signal | Measured on the day of the MRI scan
  The HC and PTS-nonSA groups will show greater ventral striatum (VS), dorsal striatum (DS), and medial prefrontal cortex (mPFC) responses during the outcome phase of the trust game for 'share' versus baseline, compared to the PTS-SA group, for the real partner condition (Trust Task), but not for the risk task.
Correlations between behavior and fMRI BOLD signal | Measured on the day of the MRI scan
  Because social withdrawal will occur in response to reduced social reward value, we hypothesize that across the PTS groups, reduced VS, DS, and mPFC activity during the outcome phase of the trust game for 'share' outcomes will be associated with lower Trust Task investments, greater self-reported social anhedonia, and smaller social network size.
PACAP correlations | Measured on the day of the MRI scan
  Elevated PACAP levels will be associated with lower investments on the Trust Task; decreased social reward signals during the outcome phase for 'share' outcomes in the VS, DS, and mPFC; and smaller social network size.

SECONDARY OUTCOMES:
Mediation analysis | Measured on the day of the MRI scan
  Within the PTS groups, decreased VS, DS, and mPFC response to 'share' outcomes will mediate the relationship between social anhedonia and reduced social network size.
Functional connectivity (psychophysiological interaction) | Measured on the day of the MRI scan
  PTS individuals with higher self-reported social anhedonia and social withdrawal will show reduced VS-mPFC connectivity for social rewards on the Trust Task.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Olson, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will evaluate requests for deidentified data on a case-by-case basis.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03383536/Prot_SAP_000.pdf